CLINICAL TRIAL: NCT03173768
Title: Quasi-experimental Study Comparing Intravenous Antibiotics Prescriptions at Hospital Discharge With and Without ID Consultation
Brief Title: Appropriateness of Intravenous Antibiotics Prescriptions at Hospital Discharge
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chiang Mai University (Other)
Responsible Party: Principal Investigator, Romanee Chaiwarith, Associate Professor, Chiang Mai University
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Health Services Research
Other Study IDs: 3631
Record Dates: First submitted 2017-04-03; First posted 2017-06-02 (Actual); Last update posted 2017-06-05 (Actual); Status verified 2017-06

CONDITIONS: Anti-Infectives Adverse Reaction
Keywords: intravenous antibiotics; appropriateness; outpatient antimicrobial therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- pre-intervention period (No Intervention): The charts of patients who were prescribed intravenous antibiotics at hospital discharge were reviewed. Appropriateness of intravenous antibiotics was assessed by ID specialists.
- post-intervention period (Experimental): The intervention is the charts of patients who were prescribed intravenous antibiotics at hospital discharge by the primary team were prospectively reviewed and intervened by ID team (ID specialist approval)
  Interventions: Procedure: ID specialist approval

INTERVENTIONS:
Procedure: ID specialist approval — Appropriateness of intravenous antibiotics ordered by the primary team was assessed by ID specialist. ID fellow modified the intravenous antibiotics ordered by the primary team if those intravenous antibiotics were judged as inappropriate by ID fellow as follows: 1) discontinue intravenous antibiotics (treatment was complete), 2) switch to oral antibiotics, 3) change intravenous antibiotics to cover isolated pathogens, 4) adjust the dose of intravenous antibiotics, and 5) change the duration of intravenous antibiotics. Finally, ID specialist retrospectively assessed the appropriateness of intravenous antibiotics at hospital discharge managed by ID fellow in post-intervention period.
  Arms: post-intervention period

SUMMARY:
A quasi-experimental study was conducted among patients receiving care at the medicine units of the Maharaj Nakorn Chiang Mai Hospital to determine the appropriateness of intravenous antibiotics at hospital discharge with and without ID consultation.

DETAILED DESCRIPTION:
The pre-intervention period was started from November 1, 2015 to April 30, 2016 (6-month period), in which the intravenous antibiotics at hospital discharge were prescribed by the primary care team. The post-intervention period was started from May 1, 2016 to February 28, 2017 (10-month period), in which the intravenous antibiotics at hospital discharge were reviewed and intervened by ID team.

The appropriateness of intravenous antibiotics was assessed separately by the ID fellow and ID specialist. If disagreement occurred, the feedback to the ID fellow was performed and the decision by ID specialist was used in the final analysis of appropriateness.

In post-intervention period, ID fellow modified the intravenous antibiotics ordered by the primary team if those intravenous antibiotics were judged as inappropriate by ID fellow as follows: 1) discontinue intravenous antibiotics (treatment was complete), 2) switch to oral antibiotics, 3) change intravenous antibiotics to cover isolated pathogens, 4) adjust the dose of intravenous antibiotics, and 5) change the duration of intravenous antibiotics

Finally, ID specialist retrospectively assessed the appropriateness of intravenous antibiotics at hospital discharge managed by ID fellow in post-intervention period.

ELIGIBILITY:
Inclusion Criteria:

All adult patients who met the following criteria were consecutively enrolled;

1. age≥ 15 years old and
2. had infections at any sites and received intravenous antibiotics.

Exclusion Criteria:

- They were evaluated by infectious diseases specialist for appropriate antibiotics during admission

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 173 (Actual)
Dates: Start 2015-11-01 (Actual); Primary Completion 2017-02-28 (Actual); Study Completion 2017-02-28 (Actual)

PRIMARY OUTCOMES:
The proportion of appropriateness of intravenous antibiotics prescriptions at hospital discharge between groups | 16 months
  To calculate the number of antibiotic prescriptions at hospital discharge over the total number of prescriptions, comparing between pre-and post-intervention period.

SECONDARY OUTCOMES:
The costs of antibiotics for the course of treatment | 16 months
  To compare the cost of antibiotics for the course of treatment between the 2 periods
Clinical improvement at 1 week | 1 week
  To calculate the number of patients who had clinical improvement at 1 week over the total number of patients in each period, comparing between the 2 periods
Readmission within 30 days, length of hospital stay | 30 days
  To calculate the number of patients who were readmitted within 30 days over the total number of patients in each period, comparing between the 2 periods
Length of hospital stay | 60 days
  To calculate the length of hospital stays in days between 2 periods

CONTACTS AND LOCATIONS:
Overall Officials: Romanee Chaiwarith, MD, Principal Investigator — Maharaj Nakorn Chiang Mai Hospital
Locations (1):
- Department of Medicine, Chiang Mai, Thailand

IPD SHARING:
Plan to Share IPD: No